CLINICAL TRIAL: NCT02292433
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, 3- Period, Crossover Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Two Dose Levels of Pf-04937319 In Japanese Subjects With Type 2 Diabetes Mellitus as Monotherapy
Brief Title: A Phase 1 Study In Japanese Subjects With Type 2 Diabetes Mellitus As Monotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B1621018
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Phase 1; type 2 diabetes; monotherapy; PF-04937319
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N,N-dimethyl-5-((2-methyl-6-((5-methylpyrazin-2-yl)carbamoyl)benzofuran-4-yl)oxy)pyrimidine-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04937319 (Experimental): PF-04937319 Split dose
  Interventions: Drug: PF-04937319 high dose; Drug: PF-04937319 low dose
- Placebo (Placebo Comparator): Placebo split dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04937319 high dose — tablets, 150 mg with breakfast plus 100 mg with lunch, 7 days
  Arms: PF-04937319
Drug: PF-04937319 low dose — tablets, 50 mg with breakfast plus 50 mg with lunch, 7 days
  Arms: PF-04937319
Drug: Placebo — tablets, breakfast plus lunch, 7 days
  Arms: Placebo

SUMMARY:
Study B1621018 will assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Two Dose Levels of Pf-04937319 in Japanese Subjects with Type 2 Diabetes Mellitus As Monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes, on diet/exercise therapy only or background therapy with 1 oral anti-diabetic agent (excluding Actos)

Exclusion Criteria:

* Patients with cardiovascular event
* Patients with diabetic complications
* Female subjects who are pregnant or planning to become pregnant
* Subjects with unstable medical conditions (eg, hypertension)

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- P-one Clinic, Keikokai Medical Corporation, Hachioji-shi, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1621018&StudyName=A%20Phase%201%20study%20in%20Japanese%20Patients%20with%20Type%202%20Diabetes%20Mellitus%20As%20Monotherapy%20

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04937319 100 mg Then PF-04937319 250 mg Then Placebo: Participants received PF-04937319 100 milligram (mg) orally per day in 2 divided doses (split dose regimen of 50 mg with morning meal and 50 mg with afternoon meal at approximately 5 hours of interval) for 7 days in the first intervention period followed by PF-04937319 250 mg orally per day in 2 divided doses (split dose regimen of 150 mg with morning meal and 100 mg with afternoon meal at approximately 5 hours of interval) for 7 days in the second intervention period, and then placebo matched to PF-04937319 administered orally with morning and afternoon meals for 7 days in the third intervention period. A washout period of 7 to 14 days was maintained between each intervention.
- PF-04937319 100 mg Then Placebo Then PF-04937319 250 mg: Participants received PF-04937319 100 mg orally per day in 2 divided doses (split dose regimen of 50 mg with morning meal and 50 mg with afternoon meal at approximately 5 hours of interval) for 7 days in the first intervention period followed by placebo matched to PF-04937319 administered orally with morning and afternoon meals for 7 days in the second intervention period, and then PF-04937319 250 mg orally per day in 2 divided doses (split dose regimen of 150 mg with morning meal and 100 mg with afternoon meal at approximately 5 hours of interval) for 7 days in the third intervention period. A washout period of 7 to 14 days was maintained between each intervention.
- Placebo Then PF-04937319 100 mg Then PF-04937319 250 mg: Participants received placebo matched to PF-04937319 administered orally with morning and afternoon meals for 7 days in the first intervention period followed by PF-04937319 100 mg orally per day in 2 divided doses (split dose regimen of 50 mg with morning meal and 50 mg with afternoon meal at approximately 5 hours of interval) for 7 days in the second intervention period, and then PF-04937319 250 mg orally per day in 2 divided doses (split dose regimen of 150 mg with morning meal and 100 mg with afternoon meal at approximately 5 hours of interval) for 7 days in the third intervention period. A washout period of 7 to 14 days was maintained between each intervention.
Period: First Intervention Period (7 Days)
Arm/Group | PF-04937319 100 mg Then PF-04937319 250 mg Then Placebo | PF-04937319 100 mg Then Placebo Then PF-04937319 250 mg | Placebo Then PF-04937319 100 mg Then PF-04937319 250 mg
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: First Washout Period (7 to 14 Days)
Arm/Group | PF-04937319 100 mg Then PF-04937319 250 mg Then Placebo | PF-04937319 100 mg Then Placebo Then PF-04937319 250 mg | Placebo Then PF-04937319 100 mg Then PF-04937319 250 mg
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Second Intervention Period (7 Days)
Arm/Group | PF-04937319 100 mg Then PF-04937319 250 mg Then Placebo | PF-04937319 100 mg Then Placebo Then PF-04937319 250 mg | Placebo Then PF-04937319 100 mg Then PF-04937319 250 mg
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Second Washout Period (7 to 14 Days)
Arm/Group | PF-04937319 100 mg Then PF-04937319 250 mg Then Placebo | PF-04937319 100 mg Then Placebo Then PF-04937319 250 mg | Placebo Then PF-04937319 100 mg Then PF-04937319 250 mg
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Third Intervention Period (7 Days)
Arm/Group | PF-04937319 100 mg Then PF-04937319 250 mg Then Placebo | PF-04937319 100 mg Then Placebo Then PF-04937319 250 mg | Placebo Then PF-04937319 100 mg Then PF-04937319 250 mg
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study medication (including placebo) in at least 1 period.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04937319 100 mg Then PF-04937319 250 mg Then Placebo | PF-04937319 100 mg Then Placebo Then PF-04937319 250 mg | Placebo Then PF-04937319 100 mg Then PF-04937319 250 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (6.6) | 52.5 (10.5) | 53.8 (6.2) | 51.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 14 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to 14 days after the last dose of study drug (minimum 8 weeks to maximum of 17 weeks)
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- PF--04937319 100 mg: All participants who received PF-04937319 100 mg orally per day in 2 divided doses (split dose regimen of 50 mg with morning meal and 50 mg with afternoon meal at approximately 5 hours of interval) for 7 days in either first or second intervention period.
- PF--04937319 250 mg: All participants who received PF-04937319 250 mg orally per day in 2 divided doses (split dose regimen of 150 mg with morning meal and 100 mg with afternoon at approximately 5 hours of interval) for 7 days in either second or third intervention period.
- Placebo: All participants who received placebo matched to PF-04937319 administered orally with morning meal and with afternoon meal for 7 days in either first, second or third intervention period.
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
participants
  AEs | 1 | 6 | 1
  SAEs | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Protocol Defined Hypoglycaemic Adverse Events (HAEs)
Description: A hypoglycemic event (HAE) was identified by characteristic symptoms or blood glucose levels. HAE was defined as 1 of the given definitions: 1) Characteristic symptoms of HAE with no home glucose monitoring performed where clinical picture included prompt resolution with food intake, subcutaneous glucagon, or intravenous glucose; 2) Characteristic symptoms of HAE with home glucose monitoring measurement of less than or equal to (=<) 70 milligram per deciliter (mg/dL) using sponsor-provided, plasma-referenced, home glucometers (or central laboratory); 3) any glucose value =<49 mg/dL using sponsor-provided, plasma-referenced, home glucometers (or central laboratory) with or without accompanying symptoms.
Time Frame: Baseline up to 14 days after the last dose of study drug (minimum 8 weeks to maximum of 17 weeks)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
participants | 1 | 4 | 0

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 1 for PF-04937319
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 1
Population: Pharmacokinetic (PK) parameter analysis population included all randomized participants who received at least 1 dose of PF-04937319 and who had at least 1 of PK parameters of interest calculated and available in at least 1 period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
nanogram per milliliter (ng/mL) | 345.8 (13) | 614.6 (20)

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 1 for PF-04937319
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 1
Population: PK parameter analysis population included all randomized participants who received at least 1 dose of PF-04937319 and who had at least 1 of PK parameters of interest calculated and available in at least 1 period.
Measure: Median (Full Range); unit: hour
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
hour | 6.50 (13) [6.50 to 6.50] | 6.50 (20) [6.50 to 8.00]

5. Primary Outcome: Area Under the Concentration-Time Curve (AUC24) From Time Zero to 24 Hour on Day 1 for PF-04937319
Description: AUC24 is the area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours post-dose (0 to 24).
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post-dose on Day 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 3308 (16) [6.50 to 6.50] | 6379 (22) [6.50 to 8.00]

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 7 for PF-04937319
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24, 36, 48 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 361.3 (16) | 692.0 (22)

7. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 7 for PF-04937319
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24, 36, 48 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
hour | 6.50 (13) [6.50 to 8.00] | 6.50 (20) [1.50 to 8.00]

8. Primary Outcome: Area Under the Concentration-Time Curve (AUC24) From Time Zero to 24 Hour on Day 7 for PF-04937319
Description: as for outcome 5
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 3840 (21) [6.50 to 6.50] | 7937 (27) [6.50 to 8.00]

9. Primary Outcome: Pre-dose Plasma Concentration (Ctrough) on Day 7 for PF-04937319
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: 0 hour (pre-dose) on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 44.82 (30) [6.50 to 6.50] | 106.3 (29) [6.50 to 8.00]

10. Primary Outcome: Average Plasma Concentration (Cav) on Day 7 for PF-04937319
Description: Cav is the average plasma concentration during the 0 to 24 hour time period.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 159.9 (21) [6.50 to 6.50] | 330.6 (27) [6.50 to 8.00]

11. Primary Outcome: Apparent Oral Clearance on Day 7 for PF-04937319
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the oral bioavailability. It is calculated as the total oral daily dose divided by AUC24, where AUC24 is the area under the plasma concentration-time profile from time 0 to 24 hours.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute (mL/min)
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
milliliter per minute (mL/min) | 434.0 (21) [6.50 to 6.50] | 525.0 (27) [6.50 to 8.00]

12. Primary Outcome: Terminal Half-Life (t1/2) on Day 7 for PF-04937319
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half. Terminal half-life is calculated by dividing the natural logarithm to the base e (Log e) multiplied by (*) 2/k el, where 'k el' is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24, 36, 48 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
hour | 8.006 (3.5291) [6.50 to 6.50] | 10.01 (4.5216) [6.50 to 8.00]

13. Primary Outcome: Apparent Volume of Distribution on Day 7 for PF-04937319
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose is influenced by the oral bioavailability. It is calculated as the total oral daily dose divided by AUC24* k el, where AUC24 is the area under the plasma concentration-time profile from time 0 to 24 hours and terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
liter | 280.5 (48) [6.50 to 6.50] | 414.6 (40) [6.50 to 8.00]

14. Primary Outcome: Accumulation Ratio (Rac) on Day 7 for PF-04937319
Description: Rac is based on AUC24. It is the ratio of AUC24 of Day 7 and AUC24 of Day 1, where AUC24 is the area under the plasma concentration-time profile from time 0 to 24 hours.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ratio | 1.159 (16) [6.50 to 6.50] | 1.244 (19) [6.50 to 8.00]

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 1 for PF-06455349
Description: PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 310.5 (21) | 583.7 (22)

16. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 1 for PF-06455349
Description: PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
hour | 11.0 (13) [11.0 to 14.0] | 11.0 (20) [8.00 to 12.5]

17. Secondary Outcome: Area Under the Concentration-Time Curve (AUC24) From Time Zero to 24 Hour on Day 1 for PF--06455349
Description: AUC24 is the area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours post-dose (0 to 24). PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 5326 (18) [6.50 to 6.50] | 10180 (19) [6.50 to 8.00]

18. Secondary Outcome: Metabolite to Parent Ratio for AUC24 (MRAUC24) on Day 1
Description: MRAUC24 is the ratio of AUC24 of PF-06455349 (metabolite) to AUC24 of PF-04937319 (parent drug) * ratio of molecular weight of PF-04937319 to molecular weight of PF-06455349, where AUC24 is the area under the plasma concentration-time profile from time 0 to 24 hours.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ratio | 1.664 (24) [6.50 to 6.50] | 1.649 (23) [6.50 to 8.00]

19. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 7 for PF--06455349
Description: PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24, 36, 48 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 464.0 (9) | 978.6 (17)

20. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 7 for PF-06455349
Description: PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24, 36, 48 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
hour | 11.0 (13) [6.50 to 12.5] | 11.0 (20) [6.50 to 12.5]

21. Secondary Outcome: Area Under the Concentration-Time Curve (AUC24) From Time Zero to 24 Hour on Day 7 for PF--06455349
Description: as for outcome 17
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 9346 (11) [6.50 to 6.50] | 19380 (15) [6.50 to 8.00]

22. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) on Day 7 for PF--06455349
Description: Ctrough is the concentration prior to study drug administration. PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose) on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 321.8 (15) [6.50 to 12.5] | 649.9 (15) [6.50 to 12.5]

23. Secondary Outcome: Average Plasma Concentration (Cav) on Day 7 for PF--06455349
Description: Cav is the average plasma concentration during the 0 to 24 hour time period. PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 389.5 (11) [6.50 to 6.50] | 807.0 (15) [6.50 to 8.00]

24. Secondary Outcome: Terminal Half-Life (t1/2) on Day 7 for PF-06455349
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half. Terminal half-life is calculated by dividing the natural logarithm to the base e (Log e) * 2/k el, where 'k el' is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression. PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24, 36, 48 hours post morning dose on Day 7
Population: PK parameter analysis population included all randomized participants who received at least 1 dose of PF-04937319 and who had at least 1 of PK parameters of interest calculated and available in at least 1 period. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 9 | 5
hour | 15.80 (1.9026) [13.2 to 18.6] | NA (NA) [14.1 to 17.3] — Data was not reported because as per planned analysis, the summary statistics was not assessed if data was missing for more than 50 percent of participants.

25. Secondary Outcome: Accumulation Ratio (Rac) on Day 7 for PF-06455349
Description: Rac is based on AUC24. It is the ratio of AUC24 of Day 7 and AUC24 of Day 1, where AUC24 is the area under the plasma concentration-time profile from time 0 to 24 hours. PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ratio | 1.756 (14) [6.50 to 6.50] | 1.903 (16) [6.50 to 8.00]

26. Secondary Outcome: Metabolite to Parent Ratio for AUC24 (MRAUC24) on Day 7
Description: MRAUC24 is the ratio of AUC24 of PF-06455349 (metabolite) to AUC24 of PF-04937319 (parent drug) * ratio of molecular weight of PF-04937319 to molecular weight of PF-06455349, where AUC24 is the area under the plasma concentration-time profile from time 0 to 24 hours. PF-06455349 is a metabolite of PF-04937319.
Time Frame: 0 hour (pre-dose), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 24 hours post morning dose on Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg
Number analyzed (Participants) | 12 | 12
ratio | 2.516 (22) [6.50 to 6.50] | 2.523 (27) [6.50 to 8.00]

27. Secondary Outcome: Change From Baseline in Weighted Mean Daily Glucose (WMDG) at Day 7
Description: WMDG was defined as time-weighted mean daily glucose. WMDG was calculated by as the time-weighted mean of glucose levels at actual time points for glucose sampling, for Day 0 (Baseline) and Day 7.
Time Frame: Pre-morning meal, 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 16 and 20 hours post- morning meal on Day 0; pre-morning dose, 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 16, 20 hours post-morning dose on Day 7
Population: The pharmacodynamic (PD) analysis population included all randomized participants who received at least 1 dose of study medication and had both a baseline and a post-baseline assessment for at least 1 PD parameter in at least 1 period.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
mg/dL
  Baseline | 201.31 (49.204) | 184.38 (51.844) | 190.42 (41.284)
  Change at Day 7 | -23.58 (14.833) | -28.61 (17.983) | 4.88 (18.182)
Statistical Analysis 1: Comparison: PF--04937319 100 mg vs Placebo; Analysis was done using a mixed effect model with sequence, period, dose, and baseline as fixed effects and participants within sequence as a random effect; Test type: Superiority or Other; p = 0.0032, Mixed Models Analysis; LS Mean Difference = -19.96, 90% CI 2-sided [-28.93 to -10.98], Standard Error of Mean 4.841
Statistical Analysis 2: Comparison: PF--04937319 250 mg vs Placebo; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -41.06, 90% CI 2-sided [-46.77 to -35.35], Standard Error of Mean 3.172

28. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Last Day of Treatment
Description: FPG was defined as plasma glucose measurements taken pre-breakfast, in the fasted state, and prior to dosing with study drug. Baseline was defined as the average of Hour 0 measurements taken on Day 0 and Day 1 in each intervention period. The measurement on the last day of treatment was defined as the average of Hour 0 measurements taken on Day 7 and Day 8 in each period.
Time Frame: Pre-morning meal on Day 0, pre-morning dose on Day 1, pre-morning dose on Day 7, pre-morning meal on Day 8
Population: PD analysis population included all randomized participants who received at least 1 dose of study medication and had both a baseline and a post-baseline assessment for at least 1 PD parameter in at least 1 period.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
mg/dL
  Baseline | 164.42 (32.389) | 156.96 (37.388) | 159.25 (30.716)
  Change at last day of treatment | -31.08 (14.860) | -39.33 (17.892) | -13.92 (17.142)
Statistical Analysis 1: Comparison: PF--04937319 100 mg vs Placebo; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = -12.18, 90% CI 2-sided [-17.16 to -7.21], Standard Error of Mean 2.851
Statistical Analysis 2: Comparison: PF--04937319 250 mg vs Placebo; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -25.81, 90% CI 2-sided [-30.73 to -20.88], Standard Error of Mean 2.821

29. Secondary Outcome: Change From Baseline in Pre-Meal Insulin at Day 7
Description: Time-matched change from baseline in pre-meal serum insulin on Day 7 of each period was analyzed. Pre-meal insulin levels therefore, pre-breakfast, pre-lunch, and pre-dinner were analyzed.
Time Frame: Pre-morning meal (pre-breakfast), 5 hours (pre-lunch), 11 hours (pre-dinner) after morning meal on Day 0 (Baseline); pre-morning dose (pre-breakfast), 5 hours (pre-lunch), 11 hours (pre-dinner) post-morning dose on Day 7
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: micro international unit per milliliter
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
micro international unit per milliliter
  Pre-breakfast: Baseline | 8.577 (4.8132) | 9.038 (5.4983) | 8.378 (5.1908)
  Pre-breakfast: Change at Day 7 | -0.828 (1.2970) | -1.439 (1.5490) | 0.594 (1.8753)
  Pre-lunch: Baseline | 10.548 (4.5632) | 9.093 (4.6060) | 9.781 (5.5415)
  Pre-lunch: Change at Day 7 | 4.258 (7.1120) | 2.640 (2.8358) | 5.416 (5.6758)
  Pre-dinner: Baseline | 13.113 (6.1401) | 13.031 (7.0380) | 13.344 (9.6188)
  Pre-dinner: Change at Day 7 | -1.625 (3.0286) | -2.521 (2.8025) | 0.449 (4.9616)
Statistical Analysis 1: Comparison: PF--04937319 100 mg vs Placebo; Analysis for pre-breakfast. Analysis was done using a mixed effect model with sequence, period, dose, and baseline as fixed effects and participants within sequence as a random effect; Test type: Superiority or Other; p = 0.0447, Mixed Models Analysis; LS Mean Difference = -1.521, 90% CI 2-sided [-2.752 to -0.290], Standard Error of Mean 0.7237
Statistical Analysis 2: Comparison: PF--04937319 250 mg vs Placebo; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.0119, Mixed Models Analysis; LS Mean Difference = -1.949, 90% CI 2-sided [-3.183 to -0.716], Standard Error of Mean 0.7249
Statistical Analysis 3: Comparison: PF--04937319 100 mg vs Placebo; Analysis for pre-lunch. Analysis was done using a mixed effect model with sequence, period, dose, and baseline as fixed effects and participants within sequence as a random effect; Test type: Superiority or Other; p = 0.6873, Mixed Models Analysis; LS Mean Difference = -0.967, 90% CI 2-sided [-5.195 to 3.261], Standard Error of Mean 2.3324
Statistical Analysis 4: Comparison: PF--04937319 250 mg vs Placebo; [analysis description as in outcome 29, analysis 3]; Test type: Superiority or Other; p = 0.0659, Mixed Models Analysis; LS Mean Difference = -2.439, 90% CI 2-sided [-4.502 to -0.377], Standard Error of Mean 0.9533
Statistical Analysis 5: Comparison: PF--04937319 100 mg vs Placebo; Analysis for pre-dinner. Analysis was done using a mixed effect model with sequence, period, dose, and baseline as fixed effects and participants within sequence as a random effect; Test type: Superiority or Other; p = 0.4031, Mixed Models Analysis; LS Mean Difference = -1.358, 90% CI 2-sided [-4.079 to 1.363], Standard Error of Mean 1.5994
Statistical Analysis 6: Comparison: PF--04937319 250 mg vs Placebo; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.0254, Mixed Models Analysis; LS Mean Difference = -3.766, 90% CI 2-sided [-6.479 to -1.052], Standard Error of Mean 1.5951

30. Secondary Outcome: Change From Baseline in Pre-Meal C-Peptide at Day 7
Description: Time-matched change from baseline in pre-meal serum C-peptide on Day 7 of each period was analyzed. Pre-meal C-peptide levels therefore, pre-breakfast, pre-lunch, and pre-dinner were analyzed.
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
ng/mL
  Pre-breakfast: Baseline | 1.68 (0.432) | 1.90 (0.663) | 1.73 (0.475)
  Pre-breakfast: Change at Day 7 | -0.38 (0.374) | -0.38 (0.325) | -0.14 (0.358)
  Pre-lunch: Baseline | 2.35 (0.674) | 2.18 (0.666) | 2.28 (0.845)
  Pre-lunch: Change at Day 7 | 0.65 (0.521) | 0.97 (0.676) | 0.84 (0.904)
  Pre-dinner: Baseline | 2.93 (0.713) | 2.93 (0.936) | 2.77 (0.951)
  Pre-dinner: Change at Day 7 | -0.64 (0.462) | -0.52 (1.079) | -0.16 (0.608)
Statistical Analysis 1: Comparison: PF--04937319 100 mg vs Placebo; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.0067, Mixed Models Analysis; LS Mean Difference = -0.21, 90% CI 2-sided [-0.33 to -0.09], Standard Error of Mean 0.069
Statistical Analysis 2: Comparison: PF--04937319 250 mg vs Placebo; [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; p = 0.0282, Mixed Models Analysis; LS Mean Difference = -0.17, 90% CI 2-sided [-0.29 to -0.05], Standard Error of Mean 0.071
Statistical Analysis 3: Comparison: PF--04937319 100 mg vs Placebo; [analysis description as in outcome 29, analysis 3]; Test type: Superiority or Other; p = 0.7877, Mixed Models Analysis; LS Mean Difference = 0.03, 90% CI 2-sided [-0.18 to 0.25], Standard Error of Mean 0.118
Statistical Analysis 4: Comparison: PF--04937319 250 mg vs Placebo; [analysis description as in outcome 29, analysis 3]; Test type: Superiority or Other; p = 0.5064, Mixed Models Analysis; LS Mean Difference = 0.11, 90% CI 2-sided [-0.17 to 0.39], Standard Error of Mean 0.156
Statistical Analysis 5: Comparison: PF--04937319 100 mg vs Placebo; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.4072, Mixed Models Analysis; LS Mean Difference = -0.25, 90% CI 2-sided [-0.75 to 0.25], Standard Error of Mean 0.293
Statistical Analysis 6: Comparison: PF--04937319 250 mg vs Placebo; [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; p = 0.1422, Mixed Models Analysis; LS Mean Difference = -0.45, 90% CI 2-sided [-0.95 to 0.06], Standard Error of Mean 0.295

ADVERSE EVENTS:
Arm/Group | PF--04937319 100 mg | PF--04937319 250 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 6/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF--04937319 100 mg (N=12) | PF--04937319 250 mg (N=12) | Placebo (N=12)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.